CLINICAL TRIAL: NCT03884998
Title: A Phase I Study of PI3Kα,δ Inhibitor Copanlisib in Combination With PD-1 Antagonist Nivolumab in Patients With Transformed Chronic Lymphocytic Leukemia (Richter's Transformation) or Non-Hodgkin Lymphoma
Brief Title: Copanlisib and Nivolumab in Treating Patients With Richter's Transformation or Transformed Indolent Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20066; NCI-2018-01880 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018655; 20066 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia; Diffuse Large B-Cell Lymphoma; Follicular Lymphoma; Indolent Non-Hodgkin Lymphoma; Lymphoplasmacytic Lymphoma; Marginal Zone Lymphoma; Richter Syndrome
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — copanlisib; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (copanlisib and nivolumab) (Experimental): Patients receive copanlisib IV over 60 minutes on days 1, 8, and 15 and nivolumab IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Copanlisib; Biological: Nivolumab

INTERVENTIONS:
Drug: Copanlisib — Given IV
  Other Names: BAY 80-6946; PI3K Inhibitor BAY 80-6946
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase I trial studies the best dose and how well copanlisib when given together with nivolumab works in treating patients with Richter's transformation or transformed indolent non-Hodgkin lymphoma. Copanlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving copanlisib and nivolumab may work better in treating patients with Richter's transformation or transformed non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the maximum-tolerated dose (MTD) of copanlisib administered in combination with nivolumab in patients with transformed chronic lymphocytic leukemia (CLL)/non-Hodgkin's lymphoma (NHL).

SECONDARY OBJECTIVE:

I. To evaluate the preliminary efficacy of copanlisib administered in combination with nivolumab in patients with transformed CLL/NHL.

EXPLORATORY OBJECTIVES:

I. To evaluate the T-cell repertoire and activation patterns following dual targeting of PI3K and PD-1.

II. To establish if PD-1/PD-L 1 expression correlates with response to the combination of copanlisib and nivolumab.

OUTLINE: This is a dose-escalation study of copanlisib.

Patients receive copanlisib intravenously (IV) over 60 minutes on days 1, 8, and 15 and nivolumab IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Richter syndrome (RS; transformed CLL), or indolent NHL (follicular lymphoma [FL], lymphoplasmacytic lymphoma [LPL], marginal zone lymphoma [MZL]) in transformation. Only patients who have diffuse large B-cell lymphoma (DLBCL) histology are eligible in transformation are eligible (for example, patients with transformation into Hodgkin lymphoma subtype are not eligible).
* Participants with RS must have received at least 2 cycles of prior systemic therapy for either RS or underlying CLL.
* Participants with FL and other indolent lymphomas in transformation must have underwent >= 1 prior chemo-immunotherapy regimen (e.g., rituximab/cyclophosphamide/doxorubicin/prednisone/vincristine [R-CHOP] or similar) administered for >= 2 cycles and have had either documented disease progression to the most recent treatment regimen, or refractory disease and must not be candidates for or planning to pursue autologous stem cell transplant, or must have relapsed following autologous stem cell transplant which took place at least 3 months prior to study therapy.
* Radiographically measurable lymphadenopathy (>= 1.5 cm) or measurable extra-nodal disease.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2.
* Total bilirubin =< 2 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x institutional ULN.
* Estimated creatinine clearance (CrCL) using the Cockroft-Gault equation >= 30 mL/min.
* Platelets >= 75,000/mm^3 (>= 25,000/mm^3 if due to disease involvement in the bone marrow; transfusion is not permitted to achieve this level).
* Absolute neutrophil count >= 1000/mm^3 (>= 500/mm^3 if due to disease involvement in the bone marrow).
* Female participants who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile (i.e. tubal ligation), OR
  * Participants of childbearing potential must have a negative serum beta-human chorionic gonadotropin at screening and:

    * Agree to practice 1 highly effective method and 1 additional effective (barrier) method of contraception at the same time, from the time of signing the informed consent through 1 month after the last dose of copanlisib, or 5 months after the last dose of nivolumab, whichever is later, or
    * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.).
* Male patients, even if surgically sterilized (i.e., status post-vasectomy) must:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 1 month after the last dose of copanlisib, OR
  * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together.).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allogeneic bone marrow or organ transplant.
* Prior therapeutic intervention with any of the following:

  * Therapeutic anti-cancer antibodies within 2 weeks.
  * Radio- or toxin-immunoconjugates within 10 weeks.
  * Radiation therapy within 2 weeks.
  * All other chemotherapy within 3 weeks prior to initiation of study therapy.
  * Targeted therapy - within 6 half-lives (for example, 36 hours for ibrutinib).
* History of prior malignancy except:

  * Malignancy treated with curative intent and no known active disease present for >= 2 years prior to initiation of therapy on current study.
  * Adequately treated non-melanoma skin cancer or lentigo maligna (melanoma in situ) without evidence of disease.
  * Adequately treated in situ carcinomas (e.g., cervical, esophageal, etc.) without evidence of disease.
  * Asymptomatic prostate cancer managed with "watch and wait" strategy.
* Any adverse event related to prior therapy that has not recovered to =< grade 1 (excluding grade 2 alopecia and grade 2 neuropathy).
* Chronic use of corticosteroids in doses which exceed 15 mg of prednisone per day, or the equivalent.
* Uncontrolled immune hemolysis or thrombocytopenia.
* A history of human immunodeficiency virus (HIV) infection. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with copanlisib and/or nivolumab. In addition, these participants are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Major surgery (under general anesthesia) within 30 days prior to therapy.
* Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV), or history of HCV.
* Live vaccine within 30 days.
* Prior PD1, PD-L 1 or checkpoint inhibitors including CTLA4, Lag3, 41BB etc. within 2 years, or at any time if administered with the intent to treat Richter syndrome.
* Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis) not requiring systemic treatment, well controlled asthma and/or mild allergic rhinitis (seasonal allergies) are eligible.
* Evidence of central nervous system (CNS) involvement.
* Use of strong CYP3A4 inhibitors or inducers within 2 weeks prior to starting study therapy.
* History or concurrent condition of interstitial lung disease and/or severely impaired lung function.
* Patients with hemoglobin (Hb) A1c > 8.5% at screening.
* Uncontrolled arterial hypertension despite optimal medical management (per investigator's assessment).
* Patients with uncontrolled coagulopathy or bleeding disorder.
* The following cardiovascular abnormalities:

  * Congestive heart failure >= class 3 New York Heart Association (NYHA) class.
  * Unstable angina (angina symptoms at rest), new-onset angina (onset within the last 3 months).
  * Myocardial infarction less than 6 months before start of study treatment.
  * Left ventricular ejection fraction (LVEF) less than 45%.
  * Corrected QT interval (QTc) > 480 msec (if echocardiogram performed during screening).
* Females who are pregnant or nursing. Pregnant individuals are excluded from this study because copanlisib and nivolumab have the potential to cause fetal harm based on relevant animal studies (Refer to the appropriate prescribing information). Because there is an unknown but potential risk for adverse events in nursing infants, breast-/chest-feeding should be discontinued prior to treatment with copanlisib and nivolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2026-11-04 (Estimated); Study Completion 2026-11-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities of copanlisib in combination with nivolumab | Up to day 28
  Will be summarized for the safety population by dose level. All adverse events (AEs) will be coded by system organ class, Medical Dictionary for Regulatory Activities (MedDRA) preferred term, and severity grade using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.
Incidence of adverse events | Up to 48 weeks
  Will be assessed by CTCAE v5. All adverse events will be tabulated and summarized by major organ category, grade, anticipation, and drug attribution. Serious adverse events (SAE) specific incidence and exact 95% confidence interval will be provided where appropriate.

SECONDARY OUTCOMES:
Overall response rate (ORR) or complete response (CR) + partial response (PR) | Up to 48 weeks
  Will be summarized with 95% confidence intervals.
Duration of response | Up to 48 weeks
  Will be summarized descriptively using means and standard deviation along with 95% confidence interval.
Progression-free survival (PFS) | Up to 48 weeks
  Will be summarized descriptively using the Kaplan-Meier estimate along with 95% confidence interval. We will also perform subset analysis with subjects who were treated at the maximum tolerated dose (MTD).

OTHER OUTCOMES:
Tumor response | Up to 48 weeks
  Will explore the association between tumor PD-L1 expression.
Evaluation of T-cell repertoire of patients with transformed chronic lymphocytic leukemia (CLL)/non-Hodgkin's lymphoma (NHL) after receiving nivolumab | Up to 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexey V Danilov, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - OHSU Knight Cancer Institute, Portland, Oregon